CLINICAL TRIAL: NCT03046121
Title: Reducing Disability Via a Family-centered Intervention for Acutely-ill Persons With Alzheimer's Disease and Related Dementias
Brief Title: A Family-centered Intervention for Acutely-ill Persons With Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Marie Boltz, Professor, Penn State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: R01AG054425 (NIH); R01AG054425 (NIH)
Record Dates: First submitted 2017-01-30; First posted 2017-02-08 (Estimated); Results first posted 2024-06-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-05

CONDITIONS: Alzheimer Disease
Keywords: dementia; acute care; post-acute recovery; family caregivers
MeSH Terms: conditions — Alzheimer Disease; Dementia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fam-FFC (Experimental): The intervention consists of :Component 1- Environmental and Policy Assessments; Component II- Education of Nursing Staff; Component III-Ongoing Training/Motivation of Nursing Staff. The Fam-FFC Nurse will work with the champions to mentor and motivate nursing staff to provide: (a) role modeling Fam-FFC, reinforcing performance of Fam-FFC, and brainstorming about ways to overcome challenges; (b) highlighting staff role models; Component IV Implementation of the FamPath Pathway which includes: (a) information on the admitting condition, diagnostics, treatment;(b) family/patient education; (c) transitional hand-off to post-acute providers; and (d) post-acute follow-up to provide ongoing education and modification of the function-focused care plan.
  Interventions: Behavioral: Family-centered Function-focused Care (Fam-FFC)
- Attention Control (Fam- FFC Ed-only) (No Intervention): Education of the nursing staff in participating hospital units (exactly as offered in treatment sites), and education of family caregivers about hospital orientation and reinforcement of discharge teaching (medications/treatments, medical follow-up).

INTERVENTIONS:
Behavioral: Family-centered Function-focused Care (Fam-FFC) — An educational empowerment model for family CGs that includes a care pathway, provided within a social-ecological in-patient framework promoting specialized care to patients with ADRD. The intervention creates an "enabling" milieu for the person with ADRD through environmental and policy assessment/modification, staff education, unit-based champions, and individualized goal setting that focuses on functional recovery during hospitalization and the immediate post-acute period.
  Arms: Fam-FFC

SUMMARY:
This study will address the effectiveness of Family-centered Function Focused Care (Fam-FFC). Fam-FFC is a theoretically-based approach to care in which family caregivers partner with nurses to prevent functional decline and other complications related to hospitalization in older adults with Alzheimer's disease and related dementias. A systematic care pathway promotes information-sharing and decision-making that promotes physical activity, function, and cognitive stimulation during the hospitalization and immediate post-acute period. Our goal in this work is to establish a practical and effective way to optimize function and physical activity; decrease neuropsychiatric symptoms, delirium, and depression; prevent avoidable post-acute care dependency; and prevent unnecessary rehospitalizations and long-stay nursing home admissions, while mitigating family caregiver strain and burden.

DETAILED DESCRIPTION:
Older persons with Alzheimer's disease and related dementias (ADRD) are about two times as likely to be hospitalized as their peers who are cognitively healthy. The care of hospitalized persons with ADRD has traditionally focused on the acute medical problem that led to admission with little attention paid to functional recovery. Older persons with ADRD are at greater risk for functional decline and increased care dependency after discharge due to a combination of intrinsic factors, environmental, policy, and care practices that restrict physical and cognitive activity, and limited staff knowledge of dementia care. Family caregivers (CGs) can play an important role in promoting the functional recovery of hospitalized older adults. They can provide vital information, offer motivation and support of function-focused care, and assume responsibility in varying degrees for post-acute care delivery and coordination. Family-centered FFC (Fam-FFC) incorporates an educational empowerment model for family CGs provided within a social-ecological in-patient framework promoting specialized care to patients with ADRD. The intervention creates an "enabling" milieu for the person with ADRD through environmental and policy assessment/modification, staff education, unit-based champions, and individualized goal setting that focuses on functional recovery. In this patient/family-centered care approach, nurses purposefully engage family CGs in the assessment, decision-making, care delivery and evaluation of function-focused care during hospitalization and the 60-day post-acute period. In the proposed project, we will implement Fam-FFC in a cluster randomized trial of 438 patient/CG dyads in six hospital units randomized within three hospitals (73 dyads per unit) to accomplish the following aims: Aim 1: Validate the efficacy of Fam-FFC on physical function (ADLs/ performance and physical activity), delirium occurrence and severity, neuropsychiatric symptoms, and mood; Aim 2: Evaluate the impact of Fam-FFC on family CG-centered outcomes (preparedness for caregiving, strain, burden, and desire to institutionalize); and Aim 3: Evaluate the relative costs for Fam-FFC v. control condition, and calculate health care cost (post-acute health care utilization) and total cost savings for Fam-FFC. We will also evaluate the cultural appropriateness of Fam-FCC for diverse families in our sample. Dyads will be composed of community-residing, hospitalized medical patients with very mild to moderate dementia (0.5 to 2.0 on the Clinical Dementia Rating Scale) and their CG (defined as the primary person providing oversight and support on an ongoing basis). Outcomes will be evaluated at hospital admission, within 72 hours of discharge, and two and six months post-discharge. This study will be a critical next step in delineating how to partner with family CGs to change acute care approaches provided to patients with ADRD so as to optimize function after discharge, and promote delirium abatement and well-being in these individuals. The societal implications of helping older individuals with Alzheimer's disease and related dementias avoid functional decline are enormous in terms of aging in place, quality of life, cost, and caregiver burden. The study findings will be relevant for other areas of behavior change research in acute care, specifically those related to engaging patients and families in health care planning, delivery, and evaluation.

ELIGIBILITY:
Patient Inclusion Criteria: medical patients who: are age ≥65, speak English or Spanish, live in the community prior to admission to the hospital, screen positive for dementia on well-validated scales (Montreal Cognitive Assessment {MoCA} ≤ 25 123-127 and AD8 >2 128,129), and score 0.5 to 2.0 on the Clinical Dementia Rating Scale; and have a family CG as the designated study partner for the duration of the study.

Patient Exclusion Criteria: mild cognitive impairment (CDR 0.5 without functional or ADL impairments), severe dementia (CDR 3), any significant neurological condition associated with cognitive impairment other than dementia (e.g. brain tumor), a major acute psychiatric disorder, have no family caregiver to participate, are enrolled in hospice and/or have a life expectancy of six months or less, are admitted from a nursing home, or experience transfers to another unit for stays longer than 48 hours.

Family Inclusion Criteria: age 18 and above whose relatives meet inclusion criteria will be eligible if they can speak and read English or Spanish; and are related to the patient by blood, marriage, adoption, or affinity as a significant other (defined as or by the patient/legally authorized person as the primary person providing oversight and support on an ongoing basis); participate, at a minimum, in the initial assessment and development of FamPath; and able to recall at least two words on the MiniCog

Staff nurses (at the conclusion of the intervention at each site) who identify the intervention unit as the primary unit worked, and speak English or Spanish, will be included in focus groups

For the exploratory aim of assessing the cultural appropriateness of the intervention, we will recruit family caregivers who self-identify as black, Latino, Asian and white, randomly selected from the Fam-FFC sample. Approximately 10 percent of families from each ethnic group represented in the study will be approached for consent for participation in interviews. (If theoretical saturation is not reached, interviews will continue until saturation is reached). Additionally, the six nurse champions will be consented and interviewed after the study ends in his/her particular unit/setting to provide their perspective on the cultural appropriateness of Fam-FFC.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 461 (Actual)
Dates: Start 2017-11-06 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2023-12-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marie Boltz, PhD, Principal Investigator — Penn State University
Locations (3):
- United States (3):
  - Lancaster General Medical Center, Lancaster, Pennsylvania
  - Presbyterian Medical Center, Philadelphia, Pennsylvania
  - Chester County Hospital, West Chester, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kuzmik A, Best I, Al Harrasi AM, Boltz M. Mediating role of care partner burden among dementia care partners during post-hospital transition. Aging Ment Health. 2024 Dec;28(12):1753-1759. doi: 10.1080/13607863.2024.2370441. Epub 2024 Jun 25. PMID 38915264
- [Derived] Kuzmik A, BeLue R, Resnick B, Rodriguez M, Berish D, Galvin JE, Boltz M. Caregiver preparedness is associated with desire to seek long-term care admission of hospitalized persons with dementia. Int J Geriatr Psychiatry. 2023 Sep;38(9):e6006. doi: 10.1002/gps.6006. PMID 37715936
- [Derived] Paudel A, Ann Mogle J, Kuzmik A, Resnick B, BeLue R, Galik E, Liu W, Behrens L, Jao YL, Boltz M. Gender differences in interactions and depressive symptoms among hospitalized older patients living with dementia. J Women Aging. 2023 Sep-Oct;35(5):476-486. doi: 10.1080/08952841.2022.2146972. Epub 2022 Nov 26. PMID 36433792
- [Derived] Boltz M, Kuzmik A, Resnick B, Trotta R, Mogle J, BeLue R, Leslie D, Galvin JE. Reducing disability via a family centered intervention for acutely ill persons with Alzheimer's disease and related dementias: protocol of a cluster-randomized controlled trial (Fam-FFC study). Trials. 2018 Sep 17;19(1):496. doi: 10.1186/s13063-018-2875-1. PMID 30223870

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was conducted between November 2017-July 2021 in six medical units across three hospitals.
Units Other Than Participants: hospital units
Period: Overall Study
Arm/Group | Fam-FFC | Attention Control (Fam- FFC Ed-only)
Started | 229; 3 hospital units | 232; 3 hospital units
Hospital 1 | 89; 1 hospital units (89 patients and 89 caregivers) | 86; 1 hospital units (86 patients and 86 caregivers)
Hospital 2 | 73; 1 hospital units (73 patients and 73 caregivers) | 73; 1 hospital units (73 patients and 73 caregivers)
Hospital 3 | 67; 1 hospital units (67 patients and 67 caregivers) | 73; 1 hospital units (73 patients and 73 caregivers)
Completed | 183; 3 hospital units | 160; 3 hospital units
Not Completed | 46; 0 hospital units | 72; 0 hospital units
Not completed — Death | 32 | 60
Not completed — Withdrawal by Subject | 14 | 12

BASELINE CHARACTERISTICS:
Population: Overall number of baseline participants is greater than the number started in the participant flow overall number as the overall number of baseline participants includes both patients and caregivers.
Units Other Than Participants: hospital units
Groups:
- Total: Total of all reporting groups
Arm/Group | Fam-FFC | Attention Control (Fam- FFC Ed-only) | Total
Number analyzed (Participants) | 458 | 464 | 922
Number analyzed (hospital units) | 3 | 3 | 6
Age, Categorical [Count of Participants; unit: Participants] — Population: Row population differs from the overall population due to attrition, which includes participants who have died, withdrawn, or were unavailable.
  Participants
    patients: number analyzed (Participants) | 229 | 232 | 461
    patients: <=18 years | 0 | 0 | 0
    patients: Between 18 and 65 years | 0 | 0 | 0
    patients: >=65 years | 229 | 232 | 461
    caregivers: number analyzed (Participants) | 213 | 222 | 435
    caregivers: <=18 years | 0 | 0 | 0
    caregivers: Between 18 and 65 years | 127 | 120 | 247
    caregivers: >=65 years | 86 | 102 | 188
Age, Continuous [Mean (Standard Deviation); unit: years]
  patients | 82.1 (8.4) | 81.1 (8.3) | 81.5 (8.4)
  caregivers | 61.0 (14.3) | 62.6 (14.1) | 61.8 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Row population differs from the overall population due to attrition, which includes participants who have died, withdrawn, or were unavailable.
  Participants
    number analyzed (Participants) | 229 | 232 | 461
    patients: Female | 145 | 130 | 275
    patients: Male | 84 | 102 | 186
    caregivers: Female | 166 | 168 | 334
    caregivers: Male | 63 | 64 | 127
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Row population differs from the overall population due to attrition, which includes participants who have died, withdrawn, or were unavailable.
  Participants
    number analyzed (Participants) | 229 | 232 | 461
    patients: Hispanic or Latino | 8 | 5 | 13
    patients: Not Hispanic or Latino | 221 | 227 | 448
    patients: Unknown or Not Reported | 0 | 0 | 0
    caregivers: Hispanic or Latino | 10 | 7 | 17
    caregivers: Not Hispanic or Latino | 216 | 221 | 437
    caregivers: Unknown or Not Reported | 3 | 4 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Row population differs from the overall population due to attrition, which includes participants who have died, withdrawn, or were unavailable.
  Participants
    number analyzed (Participants) | 229 | 232 | 461
    patients: American Indian or Alaska Native | 0 | 0 | 0
    patients: Asian | 3 | 0 | 3
    patients: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    patients: Black or African American | 89 | 76 | 165
    patients: White | 134 | 156 | 290
    patients: More than one race | 3 | 0 | 3
    patients: Unknown or Not Reported | 0 | 0 | 0
    caregivers: American Indian or Alaska Native | 0 | 0 | 0
    caregivers: Asian | 3 | 0 | 3
    caregivers: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    caregivers: Black or African American | 85 | 69 | 154
    caregivers: White | 133 | 157 | 290
    caregivers: More than one race | 5 | 2 | 7
    caregivers: Unknown or Not Reported | 3 | 4 | 7
Marital Status [Count of Participants; unit: Participants] — Population: Row population differs from the overall population due to attrition, which includes participants who have died, withdrawn, or were unavailable.
  Participants
    number analyzed (Participants) | 229 | 232 | 461
    patients: Widowed | 96 | 98 | 194
    patients: Married | 83 | 88 | 171
    patients: Other | 50 | 46 | 96
    caregivers: Widowed | 11 | 19 | 30
    caregivers: Married | 132 | 139 | 271
    caregivers: Other | 86 | 74 | 160

OUTCOME MEASURES:

1. Primary Outcome: Return to Baseline Physical Function Based on the Barthel Index (Change From 2 Weeks Prior to Admission and Changes at Admission, Discharge, and 2 and 6 Months Post-discharge).
Description: Assessed using the Barthel Index, comparing the change from 2 weeks prior to admission to changes at admission, discharge, and 2 and 6 months post-discharge. Return to baseline physical function (yes/no) was scored as yes if the participant's functional status was the same as baseline, within five points or less than baseline, or greater than baseline. Scores ranged from 0 to 1, with higher scores representing better outcomes.
Time Frame: Change from 2 weeks prior to admission to changes at admission, discharge, and 2 and 6 months post-discharge
Measure: Mean (Standard Error); unit: units on a scale
Units Other Than Participants: hospital units
Arm/Group | Fam-FFC | Attention Control (Fam- FFC Ed-only)
Number analyzed (Participants) | 229 | 232
Number analyzed (hospital units) | 3 | 3
units on a scale
  Admission | 0.68 (0.12) | 0.76 (0.10)
  Discharge | 0.77 (0.10) | 0.73 (0.11)
  2-months post discharge | 0.77 (0.10) | 0.61 (0.13)
  6-months post-discharge | 0.66 (0.12) | 0.53 (0.14)

2. Primary Outcome: Caregiver Preparedness
Description: Assessed by the Preparedness for Caregiving Scale with scores ranging from 0 to 4 and higher scores indicating greater perceived preparedness.
Time Frame: Discharge and 2 and 6 months post-discharge
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: hospital units
Arm/Group | Fam-FFC | Attention Control (Fam- FFC Ed-only)
Number analyzed (Participants) | 229 | 232
Number analyzed (hospital units) | 3 | 3
score on a scale
  Discharge | 23.7 (6.65) | 23.9 (6.93)
  2 months post-discharge | 24.1 (6.58) | 25.0 (6.38)
  6 months post-discharge | 26.5 (6.83) | 26.2 (6.63)

3. Secondary Outcome: Delirium Severity
Description: Assessed by the Confusion Assessment Method Short Form with scores ranging from 0-7 and higher scores indicating more delirium severity.
Time Frame: Admission, Discharge, 2 and 6 months post-discharge
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: hospital units
Arm/Group | Fam-FFC | Attention Control (Fam- FFC Ed-only)
Number analyzed (Participants) | 229 | 232
Number analyzed (hospital units) | 3 | 3
score on a scale
  Admission | 1.6 (1.71) | 1.3 (1.65)
  Discharge | 1.0 (1.51) | 1.0 (1.43)
  2 month post-discharge | .98 (1.46) | 1.0 (1.44)
  6 months post-discharge | 1.1 (1.57) | 1.0 (1.46)

4. Secondary Outcome: Behavior
Description: Assessed by the Brief Neuropsychiatric Inventory with scores ranging from 0 to 36 and higher scores indicating greater behavioral and psychological symptoms of dementia.
Time Frame: Admission, Discharge, 2 and 6 months post-discharge
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: hospital units
Arm/Group | Fam-FFC | Attention Control (Fam- FFC Ed-only)
Number analyzed (Participants) | 229 | 232
Number analyzed (hospital units) | 3 | 3
score on a scale
  Admission | 8.4 (6.60) | 7.2 (5.55)
  Discharge | 6.5 (6.07) | 6.3 (5.81)
  2 months post-discharge | 5.3 (6.03) | 5.4 (5.79)
  6 months post-discharge | 5.5 (6.24) | 4.6 (5.56)

5. Secondary Outcome: Moderate Physical Activity Level
Description: Actigraphy data, measured by the MotionWatch 8, includes minutes spent in moderate activity.
Time Frame: admission, discharge, 2 and 6 months post-discharge
Measure: Mean (Standard Deviation); unit: minutes
Units Other Than Participants: hospital units
Arm/Group | Fam-FFC | Attention Control (Fam- FFC Ed-only)
Number analyzed (Participants) | 229 | 232
Number analyzed (hospital units) | 3 | 3
minutes
  Admission | 4.8 (14.11) | 8.3 (29.35)
  Discharge | 14.2 (42.20) | 19.1 (48.86)
  2 months post-discharge | 23.3 (51.65) | 29.9 (63.07)
  6 months post-discharge | 27.3 (41.86) | 24.88 (43.26)

6. Secondary Outcome: Depression
Description: Assessed by the Cornell Scale for Depression in Dementia with total scores ranging between 0 to 38 and higher scores indicate more depressive symptoms.
Time Frame: admission, discharge, 2 and 6 months post-discharge
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: hospital units
Arm/Group | Fam-FFC | Attention Control (Fam- FFC Ed-only)
Number analyzed (Participants) | 229 | 232
Number analyzed (hospital units) | 3 | 3
score on a scale
  Admission | 9.4 (6.70) | 9.0 (5.72)
  Discharge | 7.5 (6.19) | 7.4 (6.02)
  2 months post-discharge | 6.2 (6.05) | 6.6 (5.95)
  6 months post-discharge | 6.2 (6.74) | 5.01 (5.44)

7. Secondary Outcome: Caregiver Strain
Description: Assessed by the Modified Caregiver Strain Index with total scores ranging from 0 to 26 and higher scores indicating greater caregiver strain.
Time Frame: Discharge and 2 and 6 months post-discharge
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: hospital units
Arm/Group | Fam-FFC | Attention Control (Fam- FFC Ed-only)
Number analyzed (Participants) | 229 | 232
Number analyzed (hospital units) | 3 | 3
score on a scale
  Discharge | 8.1 (6.53) | 7.9 (6.63)
  2 months post-discharge | 8.1 (7.02) | 7.2 (6.90)
  6 months post-discharge | 6.9 (6.83) | 6.5 (6.32)

8. Secondary Outcome: Caregiver Burden
Description: Assessed using the Short Form Zarit Burden Interview with total scores total scores ranging from 0 to 48, with higher scores corresponding to higher levels of caregiver burden.
Time Frame: Discharge and 2 and 6 months post discharge.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: hospital units
Arm/Group | Fam-FFC | Attention Control (Fam- FFC Ed-only)
Number analyzed (Participants) | 229 | 232
Number analyzed (hospital units) | 3 | 3
score on a scale
  Discharge | 10.0 (9.02) | 9.7 (9.79)
  2 months post-discharge | 13.5 (10.05) | 12.7 (9.88)
  6 months post-discharge | 9.0 (10.64) | 7.7 (9.26)

9. Secondary Outcome: Caregiver Anxiety
Description: Assessed by the Hospital Anxiety and Depression subscale with total scores ranging from 0 to 21 and higher scores indicating greater levels of caregiver anxiety.
Time Frame: Discharge and 2 and 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fam-FFC | Attention Control (Fam- FFC Ed-only)
Number analyzed (Participants) | 229 | 232
score on a scale
  Discharge | 5.4 (4.79) | 5.2 (4.72)
  2 months post-discharge | 4.7 (4.78) | 4.5 (4.76)
  6 months post-discharge | 4.7 (4.94) | 4.3 (4.91)

10. Secondary Outcome: Falls
Description: Number of falls a week after hospital discharge and 2 and 6 months post discharge.
Time Frame: discharge and 2 and 6 months
Measure: Mean (Standard Deviation); unit: Falls
Units Other Than Participants: hospital units
Arm/Group | Fam-FFC | Attention Control (Fam- FFC Ed-only)
Number analyzed (Participants) | 229 | 232
Number analyzed (hospital units) | 3 | 3
Falls
  Discharge | .15 (.55) | .14 (.66)
  2 months post-discharge | .52 (1.52) | .41 (1.19)
  6 months post-discharge | .76 (2.71) | .57 (2.17)

11. Secondary Outcome: Hospitalizations
Description: Number of hospitalizations within a week after discharge; number of hospitalizations between discharge to 2 months post-discharge; number of hospitalizations between 2 months post-discharge and 6 months post-discharge.
Time Frame: discharge and 2 and 6 months
Measure: Mean (Standard Deviation); unit: Hospitalizations
Units Other Than Participants: hospital units
Arm/Group | Fam-FFC | Attention Control (Fam- FFC Ed-only)
Number analyzed (Participants) | 229 | 232
Number analyzed (hospital units) | 3 | 3
Hospitalizations
  Discharge | .05 (.22) | .10 (.31)
  2 months post-discharge | .33 (.73) | .41 (.98)
  6 months post-discharge | .32 (.86) | .33 (.77)

12. Secondary Outcome: Emergency Room (ER) Visits
Description: Number of ER visits within a week after discharge; number of ER visits between discharge to 2 months post-discharge; number of ER visits between 2 months post-discharge and 6 months post-discharge.
Time Frame: discharge and 2 and 6 months
Measure: Mean (Standard Deviation); unit: Emergency room visits
Units Other Than Participants: hospital units
Arm/Group | Fam-FFC | Attention Control (Fam- FFC Ed-only)
Number analyzed (Participants) | 229 | 232
Number analyzed (hospital units) | 3 | 3
Emergency room visits
  Discharge | .06 (.23) | .08 (.29)
  2 months post-discharge | .41 (.80) | .44 (1.02)
  6 months post-discharge | .46 (.97) | .35 (.71)

13. Other Pre Specified Outcome: Health Care Cost
Description: cost equals staff and research nurse time (hours worked and training time) to conduct intervention.
Time Frame: end of intervention at each study site, 12 months after enrollment initiated
Population: Only participants in the Fam-FFC intervention group were measured and analyzed (i.e., contributed data reported in the table) and were included in the overall number of participants analyzed.
Measure: Mean (Standard Deviation); unit: cost in dollars
Units Other Than Participants: hospital units
Arm/Group | Fam-FFC | Attention Control (Fam- FFC Ed-only)
Number analyzed (Participants) | 229 | 0
Number analyzed (hospital units) | 3 | 0
cost in dollars | 320 (160) |

ADVERSE EVENTS:
Time Frame: admission, discharge, and 2 and 6 months post-discharge
Description: Adverse events were not monitored/assessed in the caregiver participants
Arm/Group | Fam-FFC | Attention Control (Fam- FFC Ed-only)
All-Cause Mortality (participants affected / at risk) | 32/229 | 60/232
Serious Adverse Events (participants affected / at risk) | 0/229 | 0/232
Other Adverse Events (participants affected / at risk) | 0/229 | 0/232

LIMITATIONS AND CAVEATS:
The study was limited by geographic location and attrition due to deaths which is common in this population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-08): https://cdn.clinicaltrials.gov/large-docs/21/NCT03046121/Prot_SAP_000.pdf